CLINICAL TRIAL: NCT03810495
Title: OLANI PK/Safety Study in Healthy Volunteers
Brief Title: The O'Neil Long Acting Naltrexone Implant (OLANI) Pharmacokinetic (PK)/Safety Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Go Medical Industries Pty Ltd (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); New York State Psychiatric Institute (Other); Columbia University (Other); Clinilabs, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GM0017; UG3DA047720 (NIH); 240358 (Other: NIH ERA Human Subjects Study Number)
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Opioid Use Disorder
Keywords: naltrexone; opioids; opioid use disorder; OLANI implant
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OLANI (naltrexone implant) (Experimental): 2 OLANI containing 60% naltrexone (1.8 g total) administered one time subcutaneously
  Interventions: Drug: naltrexone implant

INTERVENTIONS:
Drug: naltrexone implant — 1.8 g implant containing 60% naltrexone
  Other Names: OLANI; O'Neil Long Acting Naltrexone Implant

SUMMARY:
This study will examine the pharmacokinetic profile and safety of the O'Neil Long Acting Naltrexone Implant (OLANI) overtime in healthy volunteers. All participants will be treated in an open label manner. No randomization will occur. It is hypothesized that the OLANI will provide sustained therapeutic doses of naltrexone (NTX) for periods up to 6 months via a single subcutaneous application of 2 OLANIs.

DETAILED DESCRIPTION:
Naltrexone (NTX) is a nonspecific pure opioid antagonist with a high affinity for the µ-opioid receptor. It blocks the effects of opioids by competitive binding at opiate receptors. NTX is used primarily in the management of opiate and alcohol dependence. It is available in the United States (US) as 2 formulations; a once daily oral formulation (Revia) and a once monthly intramuscular injection (Vivitrol). While NTX is a potent antagonist and efficiently blocks the effects of exogenous opiates such as heroin, the success of NTX for the treatment of opiate dependence has been limited by poor patient compliance. Therefore, the development of a sustained release NTX formulation (in excess of 1 month) would be of great benefit for the treatment of opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 55 years old (inclusive)
* Without The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM 5) - Substance Related Disorders classification; in sustained remission is not exclusionary
* Able and willing to comply with the requirements of the protocol
* Able and willing to provide written informed consent
* Willing to undergo a minor surgical procedure under local anesthetic to allow for investigational drug administration in the subcutaneous tissue
* BMI inclusive of 18.5 to 30.0
* Have an initial weight between 45.3 and 81.6 kilograms (inclusive)

Exclusion Criteria:

* Positive urine drug screen (UDS) at screening for illicit substances.
* Is currently on naltrexone medication.
* Has had a naltrexone implant in the past 24 months.
* Has received treatment with an extended naltrexone product (e.g. Vivitrol) in the past 12 months.
* Has a condition which requires treatment with opioid based medication.
* Has a known hypersensitivity to naltrexone.
* Has a known hypersensitivity to poly-lactic based materials e.g. biodegradable sutures, surgical implants or previous biodegradable implants.
* Has a known hypersensitivity to local anesthesia.
* Is prone to skin rashes, irritation or has a skin condition such as recurrent eczema that is likely to impact the implant site area, or as determined by the evaluating physician.
* Demonstrates any abnormal skin tissue in the proposed implantation area.
* Is pregnant or planning to be. Women need to have negative blood pregnancy test at screening. Women need to agree to practice dual contraceptives.
* Participant is breastfeeding or planning to be.
* Has a current significant neurological (including cognitive and psychiatric disorders), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological or metabolic disease unless currently controlled and stable with protocol-allowed medication 30 days prior to proposed investigational product administration.
* Any clinically important abnormal finding as determined by medical history, physical examination, ECG or clinical laboratory tests.
* Any additional condition(s) that in the investigator's opinion would prohibit the participant from completing the study or would not be in the best interest of the participant.
* Alanine aminotransferase (ALT) or aspartate transaminase (AST) > 3 times the upper end of the laboratory normal range.
* Any methadone use 14 days prior to screening, and up to Study Day 0.
* Current DSM-5 diagnosis of schizophrenia, bipolar, anxiety, or depressive disorder, confirmed by The Mini International Neuropsychiatric Interview (MINI) diagnostic interview assessment, or currently treated with medications for anxiety or depression. Past history (in remission DSM-5 classification) of anxiety or depression is not exclusionary.
* Any elevated risk for suicide measured using the Columbia Suicide Severity Rating Scale (C-SSRS), endorsing any of the items in the past month (C-SSRS, Lifetime)
* Is participating or intending to participate in any other clinical trial during the duration of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OLANI (Naltrexone Implant)
Started | 20
Completed | 17
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 5
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 24.92 (3.63)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Maintain MEC
Description: Percentage of participants who maintain naltrexone (NTX) blood levels of ≥1.33 ng/mL for ≥180 days
Time Frame: up to 540 days or until NTX blood levels become undetectable
Population: Per-Protocol Population consisted of all subjects who completed at least 75% valid PK blood samples including 2 consecutive undetectable values (defined as <0.1 ng/mL) and those without any major protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
Participants | 10

2. Secondary Outcome: Median Cmax of Naltrexone
Description: Single-dose pharmacokinetic (PK) measurement of the plasma naltrexone concentration (Cmax) after dosing on Day 1
Time Frame: pre-dose, at 3, 6, and 12 hours (± 60 minutes) after dosing; 24 and 48 hours (± 2 hours) after dosing; day 4 (± 1 day), day 8 (± 2 days); days 14, 21, 28, 35, 42, 49 and 56 (± 3 days); then every 30 days (± 10 days) up to 540 days
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
ng/mL | 17.00 [5.38 to 71.4]

3. Secondary Outcome: Tmax of Naltrexone
Description: Single-dose PK measurement of the time to reach the maximum (Tmax) naltrexone concentration after dosing on Day 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
day | 49.63 [0.47 to 268]

4. Secondary Outcome: AUC of Naltrexone
Description: Single-dose PK measurement of the area under the curve (AUC) for naltrexone after dosing on Day 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: day*ng/mL
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
day*ng/mL | 1440.5 [991.1 to 2022]

5. Secondary Outcome: Median Cmax of 6β-naltrexol
Description: Single-dose PK measurement of the peak plasma 6β-naltrexol concentration after dosing on Day 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
ng/mL | 23.45 [10.2 to 126]

6. Secondary Outcome: Median Tmax of 6β-naltrexol
Description: Single-dose PK measurement of the time to reach the maximum 6β-naltrexol concentration after dosing on Day 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
day | 49.70 [1 to 176.3]

7. Secondary Outcome: Time>Minimum Effective Concentration
Description: Time (T) naltrexone remains above the minimum effective concentration (MEC) of 1.33
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
days | 270 [56 to 360]

8. Secondary Outcome: AUC of 6β-naltrexol
Description: Single-dose PK measurement of the AUC for 6β-naltrexol concentration after dosing on Day 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Full Range); unit: day*ng/mL
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 18
day*ng/mL | 2856.50 [1484 to 4990]

9. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: Incidence and Severity of AEs
Time Frame: Up to 540 days or until NTX blood levels become undetectable
Measure: Number; unit: participants
Arm/Group | OLANI (Naltrexone Implant)
Number analyzed (Participants) | 20
participants
  Participants with at least One Treatment-Emergent Adverse Event | 19
  Implant site inflammation | 7
  Vomiting | 7
  Headache | 5
  Implant site pruritus | 4
  Nausea | 3
  Diarrhoea | 3
  Upper respiratory tract infection | 3
  Implant site pain | 2
  Back pain | 2
  Weight increased | 2

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | OLANI (Naltrexone Implant)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLANI (Naltrexone Implant) (N=20)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) — Multiple severe stab wounds to the iliac crest, mid-thorax and shoulder blade
Vomiting (Gastrointestinal disorders) | 1 (1) — Cannabinoid hyperemesis syndrome
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLANI (Naltrexone Implant) (N=20)
Vomiting (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Implant site inflammation (General disorders) | 7 (7)
Implant site pruritus (General disorders) | 4 (4)
Implant site pain (General disorders) | 2 (2)
Implant site reaction (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Bacterial vaginosis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1)
Weight increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Exploratory operation (Surgical and medical procedures) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a pilot study with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03810495/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03810495/ICF_001.pdf